CLINICAL TRIAL: NCT06243003
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of Hippocampal-avoidance Whole Brain Radiotherapy Followed by Stereotactic Radiotherapy for Extensive-stage Small Cell Lung Cancer With Baseline Brain Metastases
Brief Title: WBRT With Hippocampal-avoidance Technique Followed by SRT for Extensive-stage SCLC With Baseline Brain Metastases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLC-BRT
Record Dates: First submitted 2024-01-24; First posted 2024-02-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: SCLC,Extensive Stage; Brain Metastases
Keywords: whole brain radiotherapy (WBRT); stereotactic body radiotherapy (SBRT)
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: For ES-SCLC patients with baseline brain metastasis enrolled in this study, standard chemo-immunotherapy will be delivered every 3 weeks.
  Simulation for radiotherapy should be performed at baseline, and WBRT should be completed no later than the start of the third course of systemic treatment. The WBRT dose is 30Gy/10Fx. For patients without brain metastases within 1cm of the hippocampus, hippocampal avoidance technology should be employed. After WBRT, the treating physician will perform another simulation for subsequent SRS treatment to the brain lesions. SRS should be completed no later than the start of the fourth course of drug treatment. Specific SRS dose should be as follows: 16Gy for tumors with a diameter ≤ 2cm; 12Gy for tumors with a diameter of between 2cm and 3cm. WBRT and SRS should be performed during the interval between two systemic drug treatments, concurrent (on the same day) brain radiotherapy with chemo-immunotherapy treatment should be avoided.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA-WBRT with SRS (Experimental): hippocampal-sparing WBRT combined with SRS will be used to treat SCLC patients with baseline brain metastases during standard first-line chemotherapy combined with immunotherapy.
  Interventions: Radiation: HA-WBRT plus SBRT

INTERVENTIONS:
Radiation: HA-WBRT plus SBRT — hippocampal-avoidance whole brain radiotherapy (WBRT) followed by stereotactic body radiotherapy (SBRT)

SUMMARY:
This study aims to evaluate the safety and efficacy of hippocampal-sparing WBRT combined with SRS as first-line treatment for SCLC patients with brain metastases.

DETAILED DESCRIPTION:
At present, the standard treatment for SCLC brain metastases is whole brain radiotherapy (WBRT). However, WBRT is palliative in nature due to its low dose and poor long-term control rate of intracranial lesions. At the same time, with the advent of the era of immunotherapy, a variety of PD-1/PD-L1 monoclonal antibodies combined with chemotherapy have become the standard first-line treatment for extensive-stage SCLC(ES-SCLC). Studies have shown that the survival time of SCLC patients with brain metastases is expected to be further prolonged in the era of chemotherapy and immunotherapy. Therefore, it is particularly important to further improve the control rate of intracranial lesions.

It has been confirmed in previous studies that WBRT combined with stereotactic radiotherapy for visible intracranial lesions (SRS/SRT) can effectively improve the control rate of intracranial lesions. However, most of the previous studies of WBRT combined with SRT for brain metastases did not include or only included a very small number of patients with SCLC. Studies on thoracic radiotherapy for limited-stage small cell lung cancer have found that an increase in radiotherapy dose can significantly improve the prognosis of patients with SCLC, which was previously considered to be highly radiosensitive. It is reasonable to think that SRS combined with WBRT for SCLC brain metastases may improve the prognosis of patients.

WBRT is known to cause severe cognitive impairment, which has also led to the reluctance of some patients to undergo WBRT. In the era of chemotherapy, the NRG-CC001 study showed that Hippocampal avoidance WBRT (HA-WBRT) could better protect the cognitive function of patients without affecting the prognosis of patients. The 2022 ASTRO guidelines have clearly recommended the use of hippocampal protection techniques in WBRT. Considering the lack of previous literature on the use of SRS combined with WBRT in SCLC patients in the chemo-immunotherapy era, The aim of this study is to adopt the dose fractionation of SRS combined with WBRT, which has been proven to be safe in the treatment of brain metastases from NSCLC, and to evaluate the safety of this treatment mode in SCLC patients with brain metastases receiving standard first-line chemoimmunotherapy.

In summary, this study aims to evaluate the safety and efficacy of hippocampal-sparing WBRT combined with SRS in the first-line treatment of SCLC patients with baseline brain metastases who are suitable for SRS treatment during the standard first-line chemotherapy combined with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group(ECOG) performance status score 0-2;
2. Small cell lung cancer confirmed by histopathology or cytology;
3. Complete baseline imaging data (including brain enhanced MRI/CT, positron emission tomography(PET/CT) or chest enhanced CT+ bone scan + neck and abdomen B ultrasound /CT) should be obtained before first-line treatment;
4. Patients with initial diagnosis of ES-SCLC with brain metastases who planned to receive at least 4 cycles of standard platinum-based doublet chemotherapy combined with immunotherapy (PD-1 or PD-L1 monoclonal antibody) as first-line treatment, and who met the organ function requirements as judged by the investigator;
5. Brain metastases assessed by contrast-enhanced MRI met the criteria for SRS (less than or equal to 10 brain metastases, maximum tumor volume less than 10ml, maximum tumor diameter less than 3cm, total tumor volume less than 15ml, and no evidence of leptomeningeal metastasis).
6. No history of other malignant tumors;
7. Male/female of childbearing age agreed to use contraception (surgical ligation or oral contraceptive/intrauterine device + condom) during the trial;
8. Life expectancy ≥3 months
9. Patients must be able to understand and voluntarily sign informed consent.

Exclusion Criteria:

1. Patients with non-small cell lung cancer (NSCLC) components on baseline pathological examination;
2. Patients who had received any antitumor therapy prior to ES-SCLC diagnosis;
3. Patients with imaging evidence of leptomeningeal metastasis or suspected leptomeningeal metastasis with symptoms and signs;
4. patients unable to undergo contrast-enhanced MRI;
5. Patients with severe symptoms of brain metastases requiring emergency surgery to reduce intracranial pressure;
6. Patients who could not complete immobilization for radiotherapy or tolerate radiotherapy;
7. Symptomatic interstitial lung disease or active infectious/noninfectious pneumonia;
8. Patients requiring long-term corticosteroid or immunosuppressive therapy;
9. Patients who are allergic to PD-1 or PD-L1 monoclonal antibody immunotherapy or unable to receive immune maintenance therapy for other reasons;
10. Lactating or pregnant women;
11. The patient had severe autoimmune diseases: active inflammatory bowel disease (including Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener's granulomatosis), etc.
12. Medical examination or clinical findings or other uncontrollable conditions that the investigator considers may interfere with the results or increase the risk of treatment complications for the patient;
13. Patients with mental illness, substance abuse, or social problems that could affect adherence were excluded from enrollment after physician review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicities rate | 30 days since the final day of radiotherapy
  dose-limiting toxicities(DLTs) were assessed according to CTCAE 5.0 criteria and included the following three conditions, with the exception of asymptomatic biochemical abnormalities: (1) grade 3 toxicity lasting for more than 7 consecutive days; (2) Grade 4 toxicity excluding neutropenia and thrombocytopenia; (3) Treatment-related grade 5 adverse events could not be excluded.
1-year intracranial progression-free survival rate | one year
  1-year intracranial progression-free survival (iPFS) rate was defined as proportion of patients without intracranial disease progression or death at 1 year of follow-up

SECONDARY OUTCOMES:
overall survival | one year
  overall survival(OS) was defined as the time from the date of enrollment until death by any cause. Participants still alive at the time of data analysis were censored at the date of last follow-up.
time to intracranial progression | one year
  Time to intracranial progression was defined as the time from enrollment for treatment to the observation of progression of intracranial disease.
Changes in learning and memory function | one year
  learning and memory function was assessed at 2, 4, 6, and 12 months from the first day of radiotherapy using the Hopkins Verbal Learning Test (HVLT-R)
processing speed and executive function | one year
  processing speed and executive function was assessed at 2, 4, 6, and 12 months from the first day of radiotherapy using the trail making test (TMT-Part A, to assess processing speed, and TMT-Part B, to assess executive function).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No